CLINICAL TRIAL: NCT04277598
Title: A Randomized, Placebo-controlled, Double-blind Study to Evaluate Safety and Dose Dependent Clinical Efficacy of APO-2 at Three Different Doses in Patients With Diabetic Foot Ulcer
Brief Title: A Study to Evaluate Safety and Efficacy of APO-2 at Three Different Doses in Patients With Diabetic Foot Ulcer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aposcience AG (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MARSYAS II
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Diabetic Foot Ulcer (DFU)
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: During Safety Lead In Phase 12 patients will be randomized to one of two study arms at a ratio of 3:1 between APO-2 and placebo.
  During the Main Phase 108 patients will be randomized to one of the four study arms at a ratio of 1:1:1:1 between APO-2 (three doses) and placebo.
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Lead In Phase: APO-2: 25U/ml (Experimental): Topical administration of APO-2, 25 U/ml; Approximalety 0.5 ml per square cm wound;
  Interventions: Biological: APO-2
- Lead In Phase: Placebo (Placebo Comparator): Topical administration of placebo; Approximalety 0.5 ml per square cm wound;
  Interventions: Other: Placebo
- Main Phase: APO-2: 12.5 U/ml (Experimental): Topical administration of APO-2, 12.5 U/ml; Approximalety 0.5 ml per square cm wound;
  Interventions: Biological: APO-2
- Main Phase: APO-2: 25 U/ml (Experimental): Topical administration of APO-2, 25 U/ml; Approximalety 0.5 ml per square cm wound;
  Interventions: Biological: APO-2
- Main Phase: APO-2: 50 U/ml (Experimental): Topical administration of APO-2, 50 U/ml; Approximalety 0.5 ml per square cm wound;
  Interventions: Biological: APO-2
- Main Phase: Placebo (Placebo Comparator): Topical administration of placebo; Approximalety 0.5 ml per square cm wound;
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: APO-2 — APO-2: dose adjusted gel for topical administration.
  Arms: Lead In Phase: APO-2: 25U/ml; Main Phase: APO-2: 12.5 U/ml; Main Phase: APO-2: 25 U/ml; Main Phase: APO-2: 50 U/ml
Other: Placebo — Placebo gel for topical administration.
  Arms: Lead In Phase: Placebo; Main Phase: Placebo

SUMMARY:
The MARSYAS II study which will be conducted in patients with diabetic foot ulcer (DFU) consists of a Lead-In Phase for safety assessment of multiple doses of the biologic investigational medicinal product (IMP) APO-2 and of a Main Phase (Phase II Study) to assess the efficacy and safety of the IMP. The phase II study will be a randomized study at multiple clinical centers and it will be double-blind meaning that neither the investigator nor the treated patient know if the IMP or a placebo is applied; the study will investigate the safety and clinical efficacy of multiple dose administrations at three dose levels of APO-2 (low dose, medium dose or high dose) compared with placebo.

DETAILED DESCRIPTION:
APOSEC is a secretome released by cultured, stressed peripheral blood mononuclear cells (PBMC) in medium. Content analysis revealed that APOSEC harbors a myriad of proteins, exosomes, lipids, phospholipids, cholesterols as well as antimicrobial peptides. It was shown that the topical application of APOSEC mixed with a hydrogel, called APO-2, promotes/enhances wound healing.

The MARSYAS II main study will be a multinational, multicenter, randomized, double-blind, placebo-controlled, parallel group, dose-ranging phase II study to investigate the safety and clinical efficacy of multiple dose administrations at three dose levels of APO-2 compared with placebo in patients with diabetic foot ulcer (DFU).

The main study will be preceded by a safety lead-in period evaluating multiple dose safety (25 U/ml APO-2) in patients with DFU in a cohort of 12 patients randomized at a ratio of 3:1 between APO-2 and placebo at 2 to 4 study sites. The minimum duration of an individual patient in the safety lead-in period is 93 days (including screening), with a maximum of approximately 117 days.

In the main study 120 eligible patients will be randomized at a ratio of 1:1:1:1 between APO-2 (three doses) and placebo. Patients will be stratified by wound size (at least 20% of patients will need to have wound size > 4 square cm), and randomly assigned to 1 of 4 treatment groups (low dose [12.5 U/ml], medium dose [25 U/ml], high dose [50 U/ml] or placebo). After randomization, patients will receive IMP three times per week during the 4-week active treatment period. 0.5 ml IMP will be applied per square cm wound surface area for each dose group.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 18 and 80 years of age
2. Patients with Type I or Type II diabetes with a glycosylated hemoglobin (HbA1c) of ≤ 12 %, obtained at enrollment or within 30 days prior to study enrollment
3. Patients who have a wound defined as diabetic foot ulcer present for ≥ 4 weeks
4. Foot ulcer Wagner grade I - II or ARMSTRONG grade I-A (superficial, non-infected, non-ischemic wound not involving tendon, capsules, or bone) or II-A (non-infected, non-ischemic wound penetrating to tendon or capsule but not to the bone or joint)
5. Estimated foot ulcer surface area between ≥ 0.8 cm2 and ≤ 8 cm2 as measured at day of randomization assessed using the eKare imaging and measurement device
6. A patient with more than one diabetic foot ulcer may be included in the study but only one ulcer will be selected for the investigational treatment based on Investigator judgment as far as the ulcer meets the inclusion criteria (the largest ulcer fitting the inclusion criteria will be selected as index ulcer)
7. Wound area has not changed by more than 30 % between screening visit and randomization visit (at least 14 days)
8. Adequate arterial blood perfusion measured on the leg with treated wound (ABI [ankle brachial index] ≥0.5 [the lowest ABI measured value will be used as reference], or toe pressure > 40 mmHg, or tcPO2 > 40 mmHg) within the past 6 months including patients with mild to moderate peripheral arterial disease (Fontaine Stage I and II)
9. Patient must adhere to off-loading of the ulcer area (in mobile patients adherence to off-loading footwear during the study is mandatory)
10. Patient is able to give written informed consent prior to study start and to comply with the study requirements
11. Women of childbearing potential agree using adequate birth control methods during the study

Exclusion Criteria:

1. History of anaphylaxis, known hypersensitivity to sodium alginate, propylene glycol, methylene-blue or chicken-egg
2. Target ulcer is over a deformity (such as Charcot deformity) that interferes with off-loading based on investigator's opinion
3. Index wound duration of > 3 years without intermittent healing
4. Clinical evidence of ulcer bed infection or patients requiring intravenous (IV) antibiotics to treat the index wound infection at time of randomization
5. Current evidence of osteomyelitis, cellulitis, or other evidence of infection including pus drainage from the wound site, or documented history of osteomyelitis at the target wound location during the 8 weeks preceding the screening visit
6. Major uncontrolled medical disorder(s) such as severe uncontrolled leg edema, concurrent medication, or other issue that renders the patient unsuitable for participation in the study, including but not limited to: comorbid condition with an estimated life expectancy of ≤ 12 months, hemoglobin A1c (Hba1c) > 12 % at screening, patients on dialysis, patients with severe pulmonary (requiring home oxygen, uncontrolled COPD Gold III/ IV) or cardiovascular conditions (heart failure NYHA IV, uncontrolled hypertension systolic BP by repeated measurement > 180 mmHg)
7. Raynaud disease or any other severe peripheral microvascular disease, current diagnosis of vasculitis

7a. Patients with PAD who

* have not been assessed by vascular imaging as per standard of care or
* have acute peripheral artery occlusion of the index extremity or
* have PAD Fontaine Stage III and IV or
* have PAD with planned revascularization during the upcoming 6 months or
* had Angioplasty for re-perfusion in the lower extremity with target ulcer during 3 months preceding the screening visit

  8. Dermatologic comorbid disease (e.g. pyoderma gangrenosum, vasculopathy or vasculitic ulcers), history of Systemic Lupus Erythematosus with elevated anti-DNA antibody titers, Buerger's disease (thromboangiitis obliterans)

  9. Patient currently treated for an active malignant disease or prior diagnosis of an active malignant disease who is disease free for less than 1 year. Treatment with anticancer therapy (chemotherapy, immunotherapy, radiotherapy, targeted therapy or gene therapy) within 3 months before the first administration of investigational product or at any time during the study.

  10. Patient with history of malignancy within the wound; history of radiation therapy to the wound region

  11. Patients who have undergone wound treatments with growth factors, dermal substitutes, or other biological therapies within the last 30 days or during the study

  12. Patients who received oral or parenteral corticosteroids, immunosuppressants, or cytotoxic agents within 30 days preceding the first study drug administration, or plan to use these medications during the study period

  13. Patients who are pregnant or breastfeeding

  14. Mental condition rendering the patient (or the patient's legally acceptable representative[s]) unable to understand the nature, scope and possible consequences of the study

  15. Patients who are incarcerated, including prisoners or patients compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness

  16. Therapy with another investigational agent within thirty days of screening, or during the study

  17. Patients who are considered by the investigator to have a significant disease, which can impact the study; patients who are considered not suitable for the study by the investigator

  18. Employee at the study site, spouse/partner or relative of any study staff (e.g. investigator, sub-investigators, or study nurse) or relationship to the sponsor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2020-10-09 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Wound area reduction after 4 weeks treatment with APO-2 | week 4 post baseline
  Percentage reduction in wound area from visit 2 (baseline) at day 1 to visit 14 (end of treatment) at week 4

SECONDARY OUTCOMES:
>50 % reduction in wound area | week 4 post baseline
  Proportion of patients with >50 % reduction in wound area from day 1 (baseline) to week 4 (end of treatment)
Wound size | Day 1 and week 1,2 3,4,6,8,12 post baseline
  Wound size at day 1 and 1, 2, 3, 4, 6, 8 and 12 weeks after day 1
Proportion of patients with complete wound closure | week 4, 6, 8 and 12 post baseline
  Proportion of patients with complete wound closure during 12-week follow-up period
Time to complete wound closure | A priori specification not possible; between baseline and week 12 post baseline
  Time point at which complete wound closure is achieved
Recurrence rate of the ulcer | week 4, 6, 8 and 12 post baseline
  Recurrence rate of the ulcer during 12-week follow-up period
Clinical assessment of peripheral neuropathy | day 1 and week 4 and 12 post baseline
  Assessment of severity level of peripheral neuropathy using a 10 g monofilament (Semmes-Weinstein) and a standard 128 Hz tuning fork with scaling (0 = no sense, 8 = good sense)
Assessment of local IMP tolerability | A priori specification not possible; between baseline and week 12 post baseline
  Number of patients with local adverse events with causal relationship to study medication or serious adverse events with causal relationship to study medication
Evaluation of wound pain: visual analogue scale | day 1 and week 4,6, 8 and 12 post baseline
  Evaluation of wound pain by visual analogue scale (score of 0 cm = no pain, score of 10 cm = worst pain)
Evaluation of Quality of Life: questionnaire | day 1 and week 4 and 12 post baseline
  Evaluation of Quality of Life (QoL) using Wound QoL questionnaire. Answers to each item are coded with numbers (0='not at all' to 5='very much').

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik J Ankersmit, Univ.Prof.Dr., Study Director — Aposcience AG
Locations (14):
- Austria (6):
  - LKH-Universitätsklinikum Graz; Klinische Abteilung für Plastische, Ästhetische und Rekonstruktive Chirurgie, Graz
  - Medizinische Universität Innsbruck; Univ.-Klinik für Gefäßchirurgie, Innsbruck
  - A.ö. Krankenhaus der Elisabethinen Klagenfurt GmbH; Abteilung für Chirurgie, Klagenfurt
  - Kepler Universitätsklinikum Linz; Klinik für Dermatologie und Venerologie, Linz
  - Clinic Hietzing; Wiener Gesundheitsverbund, Vienna
  - Klinikum Wels-Grieskirchen; Abteilung für Haut- und Geschlechtskrankheiten, Wels
- Czechia (4):
  - University hospital at St. Anny; Fakultní nemocnice u sv. Anny, Brno
  - University hospital Vinohrady, Prague
  - Central military hospital - Military university hospital Prague, Prague
  - Masaryk hospital in Usti nad Labem, Ústí nad Labem
- Universitätsklinikum Essen, Klinik für Endokrinologie und Stoffwechselerkrankungen, Essen, Germany
- Poland (3):
  - NZOZ "Mikomed", Lodz
  - Podos clinic, Warsaw
  - Pracownia Badań Klinicznych Salus, Wroclaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gugerell A, Gouya-Lechner G, Hofbauer H, Laggner M, Trautinger F, Almer G, Peterbauer-Scherb A, Seibold M, Hoetzenecker W, Dreschl C, Mildner M, Ankersmit HJ. Safety and clinical efficacy of the secretome of stressed peripheral blood mononuclear cells in patients with diabetic foot ulcer-study protocol of the randomized, placebo-controlled, double-blind, multicenter, international phase II clinical trial MARSYAS II. Trials. 2021 Jan 6;22(1):10. doi: 10.1186/s13063-020-04948-1. PMID 33407796